CLINICAL TRIAL: NCT00432003
Title: Neurology: A Substudy of a Large, Simple Trial Comparing Two Strategies for Management of Anti-Retroviral Therapy (SMART) to Determine the Impact of the Strategies Upon Central and Peripheral Nervous System Function
Brief Title: Effects of Anti-HIV Therapy on Nervous System Function
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 065F; CPCRA 065F1; CPCRA 065; 10115 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; HIV; Antiretroviral Therapy, Highly Active
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to observe the way two different anti-HIV treatment strategies affect nerve and brain function in adults with HIV.

DETAILED DESCRIPTION:
AIDS dementia complex (ADC) is a condition characterized by cognitive impairment, psychomotor slowing, and behavioral change. A milder form of ADC, called HIV minor cognitive/motor disorder (MCMD), is characterized by similar symptoms but has less of an impact on daily functioning. The neurocognitive impairment that results from ADC and MCMD carries an increased risk of poor drug adherence, morbidity, and mortality. It is unclear if highly active antiretroviral therapy (HAART) is effective in preserving neurocognitive function or in preventing or treating neurocognitive impairment. Distal symmetric sensory polyneuropathy (DSPN) and nucleoside-related neuropathy are two other serious conditions that HIV patients are at high risk for. DSPN is thought to be caused by active HIV infection; nucleoside-related neuropathy is thought to be caused by mitochondrial toxicity related to the use of certain antiretrovirals. These 2 conditions may lead to severe pain and discomfort in the feet. It is unknown what connection, if any, there is between DSPN and nucleoside-related neuropathy and the use of HAART. More data are needed on the natural history of these conditions.

This trial is a substudy of a study of management of antiretroviral therapy (SMART). In the SMART study, patients will participate in one of two strategies: a drug conservation (DC) strategy and a viral suppression (VS) strategy. Participants in the DC group will stop or defer HAART, then receive episodic HAART treatment for the minimum time needed to maintain a CD4 cell count of at least 250 cells/mm3. Participants in the VS group will receive HAART to maintain a viral load as low as possible, regardless of CD4 count. The purpose of this study is to compare changes in neurocognitive functioning and peripheral neuropathy symptoms between the 2 strategies of the SMART study.

Patients will participate in this substudy and the main SMART study at the same time. Within 45 days prior to randomization into the main SMART study, participants will have baseline data collected for this substudy. This data will include peripheral neuropathy assessments, treatments for symptoms of peripheral neuropathy. At selected study sites, additional measures will assess neurocognitive function, depression, alcohol and drug use, and education. At 6 months, 12 months, and every 12 months thereafter, peripheral neuropathy symptoms and treatment for the symptoms will be assessed; a pain questionnaire will also be completed. Participants will be followed until the SMART study ends.

ELIGIBILITY:
Inclusion Criteria:

* Coenrollment in the SMART study

Exclusion Criteria:

* Unable to comply with all study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2005-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change in QNPZ-5 scores
time to development of symptomatic peripheral neuropathy
change in peripheral neuropathy symptoms

SECONDARY OUTCOMES:
Time to neurocognitive impairment
time to development of ADC, stage 2 or greater
chage in peripheral neuropathy symptoms
time to development of asymptomatic or symptomatic peripheral neuropathy
time to resolution of symptomatic peripheral neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Edwina Wright, MBBS, FRACP, Study Chair — Infectious Disease Unit, the Alfred Hospital
Locations (45):
- United States (30):
  - Castro-Mission Health Ctr. CRS, San Francisco, California
  - Kaiser Permanente of Denver CRS, Denver, Colorado
  - Univ. of Colorado Health Science Ctr. CRS, Denver, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Eastside Family Health Ctr. CRS, Denver, Colorado
  - Western Infectious Disease Consultants CRS, Wheat Ridge, Colorado
  - Washington DC VAMC, Washington Regional AIDS Program, Infectious Diseases CRS, Washington D.C., District of Columbia
  - Univ. of Florida, Div. of Infectious Diseases CRS, Jacksonville, Florida
  - Earl K. Long Med. Ctr., LSU - Mid City EIC Clinic CRS, Baton Rouge, Louisiana
  - Wayne State Univ. CRS, Detroit, Michigan
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Michigan State Univ., Infectious Disease Clinic CRS, Lansing, Michigan
  - SUNY Downstate Med. Ctr., HIV Ctr. for Women & Children CRS, Brooklyn, New York
  - Harlem Hospital Ctr./Columbia University CRS (Gordin CTU), New York, New York
  - Bronx-Lebanon Hosp. Ctr. CRS, The Bronx, New York
  - Jacobi Med. Ctr., Ambulatory Care Pavillion CRS, The Bronx, New York
  - Montefiore Med. Ctr., AIDS Ctr. CRS, The Bronx, New York
  - Bronx VAMC CRS, The Bronx, New York
  - Univ. of Oklahoma Health Sciences Ctr., Div. of Infectious Diseases CRS, Oklahoma City, Oklahoma
  - The Research & Education Group-Portland CRS, Portland, Oregon
  - Kaiser Immune Deficiency Clinic of Portland CRS, Portland, Oregon
  - Legacy Clinic Emanuel CRS, Portland, Oregon
  - Oregon Health & Sciences Univ. Internal Medicine (L-475) CRS, Portland, Oregon
  - Temple Univ. School of Medicine CRS, Philadelphia, Pennsylvania
  - MediCorp, Infectious Disease Associates CRS, Fredericksburg, Virginia
  - Vernon Harris East End Community Health Ctr. CRS, Richmond, Virginia
  - CrossOver Health Ctr. CRS, Richmond, Virginia
  - VCU Health Systems, Infectious Disease Clinic CRS, Richmond, Virginia
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia
  - Med. College of Wisconsin, Infectious Disease Clinic CRS, Milwaukee, Wisconsin
- Australia (6):
  - Burwood Road Gen. Practice CRS, Burwood, New South Wales
  - St. Vincent's Hospital CRS, Darlinghurst, New South Wales
  - Westmead Hospital CRS, Westmead, New South Wales
  - Melbourne Sexual Health Ctr. CRS, Carlton, Victoria
  - The Alfred Hosp., Clinical Research - Infectious Diseases Unit CRS, Melbourne, Victoria
  - Prahran Market Clinic CRS, Melbourne, Victoria
- Brazil (2):
  - Hosp. Universitario Prof. Edgard SantosCRS, Salvador, Estado de Bahia
  - Instituto de Infectologia Emilio Ribas CRS, São Paulo
- Canada (2):
  - Q.E. II Health Sciences Ctr., Captial District Authority, Victoria Gen. Hosp. CRS, Halifax, Nova Scotia
  - Windsor Regional Hosp., HIV Care Program CRS, Windsor, Ontario
- Thailand (5):
  - Bamrasnaradura Institute CRS, Muang, Changwat Nonthaburi
  - Chulalongkorn University Hospital CRS, Bangkok, Ratchathewi
  - Mahidol Univ., Ramathibodi Hosp., Div of Infectious Disease CRS, Bangkok, Ratchathewi
  - Sanpatong Hosp. CRS, Chiang Mai
  - Khon Kaen Univ., Srinagarind Hosp., Div. of Infectious Diseases & Tropical Medicine, Dept. of Medici, Khon Kaen

REFERENCES:
- [Background] Antunes F. Central nervous system AIDS--related diseases. Acta Neurochir (Wien). 2004 Oct;146(10):1071-4. doi: 10.1007/s00701-004-0334-0. PMID 15744843
- [Background] Morgello S, Estanislao L, Simpson D, Geraci A, DiRocco A, Gerits P, Ryan E, Yakoushina T, Khan S, Mahboob R, Naseer M, Dorfman D, Sharp V; Manhattan HIV Brain Bank. HIV-associated distal sensory polyneuropathy in the era of highly active antiretroviral therapy: the Manhattan HIV Brain Bank. Arch Neurol. 2004 Apr;61(4):546-51. doi: 10.1001/archneur.61.4.546. PMID 15096404
- [Background] Sacktor N. The epidemiology of human immunodeficiency virus-associated neurological disease in the era of highly active antiretroviral therapy. J Neurovirol. 2002 Dec;8 Suppl 2:115-21. doi: 10.1080/13550280290101094. PMID 12491162
- [Background] Verma S, Estanislao L, Simpson D. HIV-associated neuropathic pain: epidemiology, pathophysiology and management. CNS Drugs. 2005;19(4):325-34. doi: 10.2165/00023210-200519040-00005. PMID 15813646
- See also: Click here for information on CPCRA 065 — http://clinicaltrials.gov/ct/show/NCT00027352